CLINICAL TRIAL: NCT02003768
Title: The Effect of Pnemoperitoneum on Intracranial Pressure and Cerebral Oxygenation During Laparoscopic Surgery According to Anesthesia Agents: Propofol Based Total Intravenous Anesthesia vs Desflurane Anesthesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 4-2013-0626
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Optic Nerve Sheath
Keywords: pneumoperitoneum; optic nerve sheath diameter; laparoscopy; Patients; general anesthesia; diameter
MeSH Terms: conditions — Pneumoperitoneum | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIVA (Experimental): 2% Propofol (Fresofol®), Remifentanil 20mcg/cc (Ultiva®)
  Interventions: Drug: Propofol
- Des (Active Comparator): Desflurane (Suprane®), Remifentanil continuous infusion (20mcg/cc)
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — 80 patients are randomly allocated into two groups: In TIVA group, propofol based total intravenous anesthesia is used to induce and maintain anesthesia for laparoscopic cholescystectomy.
  Arms: TIVA
Drug: Desflurane — 80 patients are randomly allocated into two groups : In Des group, inhalation anesthesia using desflurane is used to induce and maintain anesthesia for laparoscopic cholescystectomy.
  Arms: Des

SUMMARY:
The pneumoperitoneum during laparoscopic surgery have the potential to cause an increase of intracranial pressure (ICP). Previous studies have proposed that ultrasonographic measurements of the optic nerve sheath diameter (ONSD) correlate with signs of increased ICP. The aim of this study is to compare the effect of pnemoperitoneum on intracranial pressure and cerebral oxygenation during laparoscopic surgery according to anesthesia agents, propofol based total intravenous anesthesia (TIVA group) and desflurane anesthesia (Des group).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-80 years of age) scheduled for laparoscopic cholecystectomy undergoing general anesthesia

Exclusion Criteria:

* Patients with previous history of neurologic disease, carotid disease, transient ischemic attack, ocular disease and ocular surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
the ultrasonographic measurement of optic nerve sheath diameter | baseline
  optic nerve sheath diameter measured by ultrasonography

REFERENCES:
- [Background] Dubost C, Le Gouez A, Jouffroy V, Roger-Christoph S, Benhamou D, Mercier FJ, Geeraerts T. Optic nerve sheath diameter used as ultrasonographic assessment of the incidence of raised intracranial pressure in preeclampsia: a pilot study. Anesthesiology. 2012 May;116(5):1066-71. doi: 10.1097/ALN.0b013e318246ea1a. PMID 22258019